CLINICAL TRIAL: NCT03588312
Title: Retrospective Analysis of Results in Children Treated by an Autologous Pericardial Patch to Repair a Hypoplastic Aortic Arch Associated to Other Congenital Heart Defects
Brief Title: Long Term Results in Hypoplastic Aortic Arch Repair in Neonates Using a Glutaraldehyde Treated Autologous Pericardial Patch
Acronym: Aortoplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2017/Cardio/AorticPlasty
Record Dates: First submitted 2018-07-04; First posted 2018-07-17 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Congenital Hypoplasia of Aortic Arch
Keywords: Aortic arch hypoplasia; Glutaraldehyde treated autologous pericardium; Single stage repair; Congenital heart defects; Newborns
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- simple heart defects: Newborns with hypoplastic aortic arch in simple congenital heart defects requiring aortoplasty
  Interventions: Procedure: Aortoplasty using autologous pericardial patch
- complex heart defects.: Newborns with hypoplastic aortic arch in complex congenital heart defects requiring aortoplasty
  Interventions: Procedure: Aortoplasty using autologous pericardial patch

INTERVENTIONS:
Procedure: Aortoplasty using autologous pericardial patch — hypoplastic aortic arch repair using a glutaraldehyde treated, autologous pericardial patch.

SUMMARY:
Hypoplastic aortic arch is a congenital heart defect that is prejudicial for the growth of newborns. It is often associated to other heart defects. Different surgical techniques exist to address this defect, but the literature is very poor with regards to the use of an autologous pericardial patch. Most use extensive dissection techniques or synthetic patches. Here investigators report institution's original approach using the newborns own pericardium for what investigators believe to be an optimal correction of the hypoplasia., with preserved growth potential.

DETAILED DESCRIPTION:
Retrospective analysis of an already well codified surgical intervention carried out in HUDERF under extra-corporeal circulation

ELIGIBILITY:
Inclusion Criteria:

* Newborns with a hypoplastic aortic arch undergoing a first intervention

Exclusion Criteria:

* none

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All newborns treated in Hopital Universitaire Des Enfants - Reine Fabiola (Brussels, Belgium) for a hypoplastic aortic arch and other congenital heart defects.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 30 days post surgery

SECONDARY OUTCOMES:
Freedom from re-intervention | Up to 18 years post initial surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium